CLINICAL TRIAL: NCT02847325
Title: A Phase 1, Randomized Double-Blind, Placebo-Controlled, Single- and Multiple-Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of AC0058TA in Healthy Male and Female Subjects
Brief Title: Study of AC0058TA in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ACEA Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC00582015-101
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AC0058TA (Experimental): Drug: 50 mg AC0058TA Drug: 100 mg AC0058TA Drug: 200 mg AC0058TA Drug: 400 mg AC0058TA
  Interventions: Drug: AC0058TA
- Placebo capsules (Placebo Comparator): Drug: Placebo capsules
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: AC0058TA — 50 mg AC0058TA 100 mg AC0058TA 200 mg AC0058TA 400 mg AC0058TA
  Other Names: AC0058
  Arms: AC0058TA
Drug: Placebo capsules — Placebo capsules
  Other Names: Placebo
  Arms: Placebo capsules

SUMMARY:
AC0058TA is a small molecule compound that potently, selectively and irreversibly inhibits Bruton's tyrosine kinase (BTK) phosphorylation and downstream signals, resulting in inhibition of inflammatory cytokine production in monocytes and inhibition of lymphocyte activation (predominantly B-cell activation) in the preclinical studies. The nonclinical program has demonstrated that AC0058TA has the potential to interfere with signaling functions mediated by tyrosine kinases and may be useful for controlling excessive or aberrant T- and B-cell activation in autoimmune diseases.

As an investigational targeted therapy for RA and SLE, AC0058TA is expected to address the unmet need of this patient population, for whom there are currently no effected therapies and there is a great unmet medical need, AC0058TA may inhibit the key pathway which involves the disease process.

DETAILED DESCRIPTION:
This is a 2-part, randomized, double-blind, placebo-controlled, single-dose-escalation (Part 1) and multiple-dose-escalation (Part 2) study to evaluate the safety, tolerability, PK, and PD of AC0058TA administered orally to healthy subjects. Part 1 of the study will also to evaluate the effect of food on the pharmacokinetics of a single oral dose of AC0058TA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any ethnic origin, age ≥18 and ≤65 years of age;
* BMI ≥18.5 and ≤32.0 kg/m2;
* Medical history without major pathology and determined to be in good health with no clinically significant findings as assessed by the Investigator;
* All clinical laboratory tests of blood and urine are within the normal range or show no clinically relevant deviations as judged by the Investigator;
* A female must be

  * postmenopausal (ie, have spontaneous amenorrhea for ≥12 consecutive months with follicle stimulating hormone (FSH) ≥40 mIU/mL at Screening, and be of an appropriate age) or
  * surgically sterile (ie, hysterectomy, bilateral salpingectomy, bilateral oophorectomy, tubal occlusion) for at least 90 days prior to Screening;
* Male subjects must agree to use at least 2 methods of contraception with a female partner of childbearing potential, with at least 1 method being a highly effective method of contraception (as defined in Section 5.5), to refrain from sperm donation, and to refrain from unprotected sexual intercourse with a female who is pregnant or breastfeeding during the study from the time of signing the informed consent or 10 days prior to Check-in (Day -1) until 90 days after the last administration of study medication or discontinuation;
* Able to comprehend and abide by the study restrictions, and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

* Has a significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, immune suppressive/defective, or psychiatric disorder as determined by the Investigator;
* Has a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;
* Has a history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (a subject who has had an appendectomy or hernia repair may be enrolled in the study);
* Has a history of congenital nonhemolytic hyperbilirubinaemia (eg, Gilbert's syndrome);
* Has a history of alcoholism or drug addiction within 1 year prior to Check-in;
* Has a positive test for selected drugs of abuse at Screening (not including alcohol) or Check-in (including alcohol);
* Has a positive hepatitis panel and/or positive human immunodeficiency virus (HIV) antibody screens;
* Has a positive pregnancy test result at Screening or Check-in (females only);
* Has clinically significant findings as determined by the Investigator (eg, medical history, 12-lead ECG, vital signs, or clinical laboratory evaluations;
* Has participated in any other investigational drug trial in which receipt of an investigational drug (new chemical entity) occurred within 5 half-lives of the respective study drug or 30 days prior to Check-in, whichever is longer;
* Has used any medications/products, including St. John's Wort, known to alter drug absorption or elimination processes within 30 days prior to Check-in, unless deemed acceptable by the Investigator;
* Has used any prescription medications/products not discussed in another exclusion criterion within 14 days prior to Check-in, unless deemed acceptable by the Investigator;
* Has used slow-release medications/products considered to still be active within 14 days prior to Check-in, unless deemed acceptable by the Investigator; 14. Has used any over-the-counter, nonprescription medications/products not discussed in another exclusion criterion (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in, unless deemed acceptable by the Investigator;
* Has donated blood within 30 days prior to Screening, plasma within 2 weeks prior to Screening, or platelets within 6 weeks prior to Screening;
* Has received blood products within 2 months prior to Check-in;
* Has poor peripheral venous access;
* Who, in the opinion of the Investigator, should not participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-05; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple oral doses of AC0058TA determined by adverse events | within 6 days after single dose in part 1, within 14 days after last dose in part 2.
  Frequency and severity of AEs and serious AEs

SECONDARY OUTCOMES:
Plasma concentrations of single dose or multiple doses of AC0058TA | within 6 days after single dose in part 1, within 14 days after last dose in part 2.
  Maximum observed concentration (Cmax)
Time to maximum observed concentration (Tmax) | within 6 days after single dose in part 1, within 14 days after last dose in part 2.
  Time to maximum observed concentration (Tmax)
Area under the concentration-time curve (AUC) | within 6 days after single dose in part 1, within 14 days after last dose in part 2.
  Area under the concentration-time curve (AUC)
The effect of food on AUC of the single-oral-dose AC0058TA | within 6 days after single dose in part 1
  Area under the concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Development Services, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided